CLINICAL TRIAL: NCT00400153
Title: Safety and Efficacy of Combivent Respimat in Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Respimat® Combivent Trial in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1012.56; NCT00847652 (obsolete NCT alias)
Record Dates: First submitted 2006-11-15; First posted 2006-11-16 (Estimated); Results first posted 2009-06-01 (Estimated); Last update posted 2014-06-13 (Estimated); Status verified 2014-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol, Ipratropium Drug Combination

ARMS (3):
- COMBIVENT Respimat 20/100 mcg (Experimental)
  Interventions: Drug: Combivent Respimat (20 mcg/100 mcg); Drug: Placebo via corresponding inhaler for blinding purposes
- COMBIVENT CFC-MDI 36/206 mcg (Experimental)
  Interventions: Drug: COMBIVENT MDI (36/206 mcg); Drug: Placebo via corresponding inhaler for blinding purposes
- Ipratropium Respimat 20 mcg (Experimental)
  Interventions: Drug: Atrovent Respimat (20 mcg); Drug: Placebo via corresponding inhaler for blinding purposes

INTERVENTIONS:
Drug: Atrovent Respimat (20 mcg)
  Arms: Ipratropium Respimat 20 mcg
Drug: COMBIVENT MDI (36/206 mcg)
  Arms: COMBIVENT CFC-MDI 36/206 mcg
Drug: Combivent Respimat (20 mcg/100 mcg)
  Arms: COMBIVENT Respimat 20/100 mcg
Drug: Placebo via corresponding inhaler for blinding purposes

SUMMARY:
The primary objective of this study is to compare the effect of ipratropium bromide/salbutamol inhalation spray combination administered by the Respimat® inhaler (20 mcg/100 mcg), ipratropium bromide inhalation spray administered by the Respimat® inhaler (20 mcg), and COMBIVENT® MDI administered q.i.d on FEV1 at intervals over a treatment period of 12 weeks in patients with COPD. Specifically, non-inferiority of Combivent Respimat® to COMBIVENT® MDI in FEV1 AUC from 0 to 6 hours , superiority of Combivent Respimat® to Atrovent Respimat® monotherapy in FEV1 AUC from 0 to 4 hours, and non-inferiority of Combivent Respimat® to Atrovent Respimat® monotherapy in FEV1 AUC from 4 to 6 hours will be analyzed. In addition, steady state pharmacokinetics over one dosing interval following 4 weeks of therapy will be characterized in a subgroup of patients.

ELIGIBILITY:
Inclusion Criteria:

Outpatients of either sex, 40 years or older, with a diagnosis of COPD (FEV1 65% predicted normal and FEV1/FVC 70%).

Exclusion Criteria:

Patients with significant diseases other than COPD that may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study, with a history of asthma or allergic rhinitis, who regularly use daytime oxygen therapy for more than 1 hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy or using oral corticosteroid me dication at unstable doses (i.e., less than 6 weeks on a stable dose) or at a dose in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day will be excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1480 (Actual)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (180):
- United States (87):
  - 1012.56.01006 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1012.56.01051 Boehringer Ingelheim Investigational Site, Jasper, Alabama
  - 1012.56.01071 Boehringer Ingelheim Investigational Site, Mobile, Alabama
  - 1012.56.01039 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1012.56.01012 Boehringer Ingelheim Investigational Site, Lakewood, California
  - 1012.56.01029 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1012.56.01043 Boehringer Ingelheim Investigational Site, Palo Alto, California
  - 1012.56.01089 Boehringer Ingelheim Investigational Site, Rancho Mirage, California
  - 1012.56.01021 Boehringer Ingelheim Investigational Site, Riverside, California
  - 1012.56.01033 Boehringer Ingelheim Investigational Site, San Jose, California
  - 1012.56.01020 Boehringer Ingelheim Investigational Site, Sepulveda, California
  - 1012.56.01045 Boehringer Ingelheim Investigational Site, Torrence, California
  - 1012.56.01040 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1012.56.01050 Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - 1012.56.01018 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1012.56.01062 Boehringer Ingelheim Investigational Site, Wheat Ridge, Colorado
  - 1012.56.01036 Boehringer Ingelheim Investigational Site, Hartford, Connecticut
  - 1012.56.01025 Boehringer Ingelheim Investigational Site, Stamford, Connecticut
  - 1012.56.01088 Boehringer Ingelheim Investigational Site, Waterbury, Connecticut
  - 1012.56.01007 Boehringer Ingelheim Investigational Site, Bay Pines, Florida
  - 1012.56.01058 Boehringer Ingelheim Investigational Site, Brandon, Florida
  - 1012.56.01010 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1012.56.01065 Boehringer Ingelheim Investigational Site, Clearwater, Florida
  - 1012.56.01024 Boehringer Ingelheim Investigational Site, DeLand, Florida
  - 1012.56.01001 Boehringer Ingelheim Investigational Site, Melbourne, Florida
  - 1012.56.01023 Boehringer Ingelheim Investigational Site, Panama City, Florida
  - 1012.56.01052 Boehringer Ingelheim Investigational Site, Pensecola, Florida
  - 1012.56.01048 Boehringer Ingelheim Investigational Site, Tampa, Florida
  - 1012.56.01093 Boehringer Ingelheim Investigational Site, Winter Park, Florida
  - 1012.56.01077 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1012.56.01083 Boehringer Ingelheim Investigational Site, Decatur, Georgia
  - 1012.56.01008 Boehringer Ingelheim Investigational Site, Coeur d'Alene, Idaho
  - 1012.56.01019 Boehringer Ingelheim Investigational Site, Olathe, Kansas
  - 1012.56.01056 Boehringer Ingelheim Investigational Site, Wichita, Kansas
  - 1012.56.01066 Boehringer Ingelheim Investigational Site, Bowling Green, Kentucky
  - 1012.56.01090 Boehringer Ingelheim Investigational Site, Lafayette, Louisiana
  - 1012.56.01054 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1012.56.01072 Boehringer Ingelheim Investigational Site, New Orleans, Louisiana
  - 1012.56.01070 Boehringer Ingelheim Investigational Site, Shreveport, Louisiana
  - 1012.56.01035 Boehringer Ingelheim Investigational Site, Baltimore, Maryland
  - 1012.56.01079 Boehringer Ingelheim Investigational Site, Ann Arbor, Michigan
  - 1012.56.01044 Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - 1012.56.01076 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1012.56.01082 Boehringer Ingelheim Investigational Site, Henderson, Nevada
  - 1012.56.01049 Boehringer Ingelheim Investigational Site, Reno, Nevada
  - 1012.56.01080 Boehringer Ingelheim Investigational Site, Brick, New Jersey
  - 1012.56.01027 Boehringer Ingelheim Investigational Site, Cherry Hill, New Jersey
  - 1012.56.01028 Boehringer Ingelheim Investigational Site, Summit, New Jersey
  - 1012.56.01069 Boehringer Ingelheim Investigational Site, Albuquerque, New Mexico
  - 1012.56.01022 Boehringer Ingelheim Investigational Site, Larchmont, New York
  - 1012.56.01015 Boehringer Ingelheim Investigational Site, New Hyde Park, New York
  - 1012.56.01068 Boehringer Ingelheim Investigational Site, New York, New York
  - 1012.56.01078 Boehringer Ingelheim Investigational Site, Asheville, North Carolina
  - 1012.56.01017 Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - 1012.56.01042 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1012.56.01034 Boehringer Ingelheim Investigational Site, Sylvania, Ohio
  - 1012.56.01031 Boehringer Ingelheim Investigational Site, Toledo, Ohio
  - 1012.56.01038 Boehringer Ingelheim Investigational Site, Oklahoma City, Oklahoma
  - 1012.56.01016 Boehringer Ingelheim Investigational Site, Medford, Oregon
  - 1012.56.01067 Boehringer Ingelheim Investigational Site, Hershey, Pennsylvania
  - 1012.56.01003 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1012.56.01060 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
  - 1012.56.01004 Boehringer Ingelheim Investigational Site, Pittsburgh, Pennsylvania
  - 1012.56.01087 Boehringer Ingelheim Investigational Site, East Providence, Rhode Island
  - 1012.56.01057 Boehringer Ingelheim Investigational Site, Johnston, Rhode Island
  - 1012.56.01026 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1012.56.01037 Boehringer Ingelheim Investigational Site, Charleston, South Carolina
  - 1012.56.01081 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1012.56.01085 Boehringer Ingelheim Investigational Site, Greenville, South Carolina
  - 1012.56.01084 Boehringer Ingelheim Investigational Site, Greer, South Carolina
  - 1012.56.01011 Boehringer Ingelheim Investigational Site, Spartanburg, South Carolina
  - 1012.56.01073 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1012.56.01075 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1012.56.01047 Boehringer Ingelheim Investigational Site, Fort Worth, Texas
  - 1012.56.01014 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1012.56.01032 Boehringer Ingelheim Investigational Site, Killeen, Texas
  - 1012.56.01002 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1012.56.01053 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1012.56.01009 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1012.56.01013 Boehringer Ingelheim Investigational Site, Richmond, Virginia
  - 1012.56.01059 Boehringer Ingelheim Investigational Site, Roanoke, Virginia
  - 1012.56.01055 Boehringer Ingelheim Investigational Site, Salem, Virginia
  - 1012.56.01063 Boehringer Ingelheim Investigational Site, Bellington, Washington
  - 1012.56.01005 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1012.56.01064 Boehringer Ingelheim Investigational Site, Spokane, Washington
  - 1012.56.01030 Boehringer Ingelheim Investigational Site, Tacoma, Washington
  - 1012.56.01074 Boehringer Ingelheim Investigational Site, Morgantown, West Virginia
- Argentina (15):
  - 1012.56.54001 Centro Médico de la Dra. De Salvo, Capital Federal
  - 1012.56.54002 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1012.56.54003 Policlínica Bancaria, Capital Federal
  - 1012.56.54004 Hospital Ramos Mejia, Capital Federal
  - 1012.56.54010 Instituto Lanari, Capital Federal
  - 1012.56.54011 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1012.56.54015 Boehringer Ingelheim Investigational Site, Capital Federal
  - 1012.56.54005 Instituto de Diagnóstico Cardiovascular La Plata, La Plata
  - 1012.56.54012 Boehringer Ingelheim Investigational Site, Lanús
  - 1012.56.54009 Instituto de Investigaciones Clínicas, Mar del Plata
  - 1012.56.54014 Boehringer Ingelheim Investigational Site, Mendoza
  - 1012.56.54007 CLINICA PRIVADA de MONTE GRANDE, Monte Grande
  - 1012.56.54006 CENTRO PRIVADO de MEDICINA RESPIRATORIA, Paraná
  - 1012.56.54008 HOSPITAL ITALIANO de ROSARIO, Rosario
  - 1012.56.54013 Boehringer Ingelheim Investigational Site, San Miguel de Tucumán
- France (6):
  - 1012.56.3305A Centre hospitalier Germon & Gauthier, Béthune
  - 1012.56.3303A Clinique de la Louvière, Lille
  - 1012.56.3301A Hôpital Ambroise Paré, Marseille
  - 1012.56.3304A Centre Médical Erdre Saint Augustin, Nantes
  - 1012.56.3302A Cabinet Médical, Nice
  - 1012.56.3302B Cabinet Médical, Nice
- Greece (9):
  - 1012.56.30001 Boehringer Ingelheim Investigational Site, Athens
  - 1012.56.30011 Boehringer Ingelheim Investigational Site, Athens
  - 1012.56.30013 Boehringer Ingelheim Investigational Site, Athens
  - 1012.56.30010 Boehringer Ingelheim Investigational Site, Corinth
  - 1012.56.30009 Boehringer Ingelheim Investigational Site, Heraklion
  - 1012.56.30007 Boehringer Ingelheim Investigational Site, Komotini
  - 1012.56.30002 Boehringer Ingelheim Investigational Site, Larissa
  - 1012.56.30014 Boehringer Ingelheim Investigational Site, Nafplion
  - 1012.56.30003 Boehringer Ingelheim Investigational Site, Thessaloniki
- New Zealand (5):
  - 1012.56.64004 Boehringer Ingelheim Investigational Site, Dunedin
  - 1012.56.64001 Boehringer Ingelheim Investigational Site, Grafton / Auckland
  - 1012.56.64003 Boehringer Ingelheim Investigational Site, Hamilton
  - 1012.56.64006 Boehringer Ingelheim Investigational Site, Tauranga
  - 1012.56.64005 Boehringer Ingelheim Investigational Site, Wellington
- Poland (10):
  - 1012.56.48009 Boehringer Ingelheim Investigational Site, Bydgoszcz
  - 1012.56.48006 Boehringer Ingelheim Investigational Site, Krakow
  - 1012.56.48007 Boehringer Ingelheim Investigational Site, Krakow
  - 1012.56.48004 Boehringer Ingelheim Investigational Site, Ostrow Wielkopolska
  - 1012.56.48005 Boehringer Ingelheim Investigational Site, Poznan
  - 1012.56.48002 Boehringer Ingelheim Investigational Site, Proszowice
  - 1012.56.48010 Boehringer Ingelheim Investigational Site, Radom
  - 1012.56.48001 Boehringer Ingelheim Investigational Site, Warsaw
  - 1012.56.48011 Boehringer Ingelheim Investigational Site, Warsaw
  - 1012.56.48003 Boehringer Ingelheim Investigational Site, Wroclaw
- Russia (8):
  - 1012.56.07010 Boehringer Ingelheim Investigational Site, Kazan'
  - 1012.56.07001 Boehringer Ingelheim Investigational Site, Moscow
  - 1012.56.07002 Boehringer Ingelheim Investigational Site, Moscow
  - 1012.56.07003 Boehringer Ingelheim Investigational Site, Moscow
  - 1012.56.07005 Boehringer Ingelheim Investigational Site, Moscow
  - 1012.56.07007 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1012.56.07008 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1012.56.07009 Boehringer Ingelheim Investigational Site, Saint Petersburg
- South Africa (8):
  - 1012.56.27002 Boehringer Ingelheim Investigational Site, Bellville
  - 1012.56.27008 Boehringer Ingelheim Investigational Site, Boksburg
  - 1012.56.27001 Boehringer Ingelheim Investigational Site, Cape Town
  - 1012.56.27004 Boehringer Ingelheim Investigational Site, Cape Town
  - 1012.56.27005 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1012.56.27009 Boehringer Ingelheim Investigational Site, Orange Grove
  - 1012.56.27003 Boehringer Ingelheim Investigational Site, Paarl
  - 1012.56.27006 Boehringer Ingelheim Investigational Site, Park Town West
- South Korea (8):
  - 1012.56.82009 Boehringer Ingelheim Investigational Site, Daegu
  - 1012.56.82010 Boehringer Ingelheim Investigational Site, Geonggi-Do
  - 1012.56.82008 Boehringer Ingelheim Investigational Site, Gyeonggi-do
  - 1012.56.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1012.56.82002 Boehringer Ingelheim Investigational Site, Seoul
  - 1012.56.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1012.56.82006 Boehringer Ingelheim Investigational Site, Seoul
  - 1012.56.82007 Boehringer Ingelheim Investigational Site, Seoul
- Taiwan (5):
  - 1012.56.88604 Chang Gong Memorial Hospital, Keelong Town
  - 1012.56.88605 Taichung Veterans General Hospital, Taichung
  - 1012.56.88602 Taipei Veterans General Hospital, Taipei
  - 1012.56.88603 National Taiwan University Hospital, Taipei
  - 1012.56.88601 Chang Gung Memorial Hosp-Linkou, Taoyuan District
- Turkey (Türkiye) (5):
  - 1012.56.90001 Boehringer Ingelheim Investigational Site, Ankara
  - 1012.56.90005 Boehringer Ingelheim Investigational Site, Antalya
  - 1012.56.90003 Boehringer Ingelheim Investigational Site, Istanbul
  - 1012.56.90006 Boehringer Ingelheim Investigational Site, Istanbul
  - 1012.56.90002 Boehringer Ingelheim Investigational Site, Mersin
- Ukraine (5):
  - 1012.56.38005 Boehringer Ingelheim Investigational Site, Dnyepropyetrovsk
  - 1012.56.38006 Boehringer Ingelheim Investigational Site, Donetsk
  - 1012.56.38001 Boehringer Ingelheim Investigational Site, Kiev
  - 1012.56.38002 Boehringer Ingelheim Investigational Site, Kiev
  - 1012.56.38004 Boehringer Ingelheim Investigational Site, Kiev
- United Kingdom (9):
  - 1012.56.44009 Boehringer Ingelheim Investigational Site, Ballieston, Glasgow
  - 1012.56.44003 Boehringer Ingelheim Investigational Site, Bury Saint Edmonds
  - 1012.56.44002 Boehringer Ingelheim Investigational Site, Cambridge
  - 1012.56.44006 Colchester General Hospital, Colchester
  - 1012.56.44007 Boehringer Ingelheim Investigational Site, Doncaster
  - 1012.56.44001 Medicine Evaluation Unit, Manchester
  - 1012.56.44008 The Staploe Medical Centre, Soham
  - 1012.56.44005 Morriston Hospital, Swansea
  - 1012.56.44010 Boehringer Ingelheim Investigational Site, Windsor

REFERENCES:
- [Derived] Zuwallack R, De Salvo MC, Kaelin T, Bateman ED, Park CS, Abrahams R, Fakih F, Sachs P, Pudi K, Zhao Y, Wood CC; Combivent Respimat Inhaler Study Group. Efficacy and safety of ipratropium bromide/albuterol delivered via Respimat inhaler versus MDI. Respir Med. 2010 Aug;104(8):1179-88. doi: 10.1016/j.rmed.2010.01.017. Epub 2010 Feb 20. PMID 20172704

RESULTS

PARTICIPANT FLOW:
Groups:
- COMBIVENT Respimat 20/100 mcg: Combivent Respimat (20 mcg/100 mcg) plus placebo COMBIVENT MDI
- COMBIVENT CFC-MDI 36/206 mcg: COMBIVENT MDI (36/206 mcg ) plus placebo Combivent Respimat
- Ipratropium Respimat 20 mcg: Atrovent Respimat (20 mcg) plus placebo COMBIVENT MDI
Period: Overall Study
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Started | 486 | 491 | 483
Completed | 438 | 436 | 422
Not Completed | 48 | 55 | 61
Not completed — AE due to study disease worsening | 14 | 19 | 20
Not completed — AE due to other disease worsening | 2 | 1 | 0
Not completed — AE due to other condition | 3 | 14 | 15
Not completed — Protocol Violation | 7 | 4 | 9
Not completed — Lost to Follow-up | 2 | 1 | 4
Not completed — Withdrawal by Subject | 12 | 11 | 10
Not completed — Other reasons - not mentioned above | 8 | 5 | 3

BASELINE CHARACTERISTICS:
Population: The treated set (TS) included all randomized patients who were documented to have taken at least one actuation of the randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg | Total
Number analyzed (Participants) | 486 | 491 | 483 | 1460
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (8.7) | 64.2 (9.2) | 64.3 (8.6) | 64.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 170 | 169 | 166 | 505
  Male | 316 | 322 | 317 | 955
Race/Ethnicity, Customized [Number; unit: participants]
  White | 430 | 442 | 428 | 1300
  Black | 27 | 25 | 26 | 78
  Asian | 29 | 24 | 29 | 82
Height [Mean (Standard Deviation); unit: cm] | 168.8 (9.1) | 169.4 (9.4) | 168.8 (9.5) | 169.3 (9.3)
Weight [Mean (Standard Deviation); unit: kg] | 78.2 (20.0) | 77.8 (19.3) | 77.3 (21.0) | 77.8 (20.1)
Alcoholic history [Number; unit: participants]
  Non drinker | 223 | 232 | 223 | 678
  Drinks - not interfere with participation in trial | 263 | 258 | 260 | 781
  Drinks-poss. interfere with participation in trial | 0 | 1 | 0 | 1
Smoking history [Mean (Standard Deviation); unit: pack years] | 51.7 (27.7) | 52.4 (27.1) | 55.4 (27.6) | 53.2 (27.5)
COPD duration [Mean (Standard Deviation); unit: years] | 8.2 (6.1) | 8.6 (6.5) | 8.5 (6.4) | 8.4 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC0-6 at Day 85
Description: Area between the test-day baseline FEV1 and the FEV1 change from the test-day baseline curve from 0 to 6 hours divided by 6 at Day 85
Time Frame: Before drug administration to 6 hours after drug administration on Day 85
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.145 (0.007) | 0.149 (0.007) | 0.119 (0.007)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.05 liter; p = 0.7135, ANCOVA; Mean Difference (Final Values) = -0.0035, 95% CI [-0.0222 to 0.0152], Standard Error of Mean 0.0095

2. Primary Outcome: FEV1 AUC0-4 at Day 85
Description: Area between the test-day baseline FEV1 and the FEV1 change from the test-day baseline curve from 0 to 4 hours divided by 4 at Day 85
Time Frame: Before drug administration to 4 hours after drug administration on Day 85
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.189 (0.007) | 0.190 (0.007) | 0.142 (0.007)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.047, 95% CI [0.028 to 0.066], Standard Error of Mean 0.01

3. Primary Outcome: FEV1 AUC4-6 at Day 85
Description: Area between the test-day baseline FEV1 and the FEV1 change from the test-day baseline curve from 4 to 6 hours divided by 2 at Day 85
Time Frame: Between 4 hours and 6 hours after drug administration on Day 85
Population: Full Analysis Set for Pulmonary Function Test Data 4-6 hours
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 447 | 449 | 427
liters | 0.056 (0.008) | 0.066 (0.008) | 0.073 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; Test type: Non-Inferiority or Equivalence — Non-inferiority margin is 0.05 liters; p = 0.1389, ANCOVA; Mean Difference (Final Values) = -0.017, 95% CI [-0.039 to 0.005], Standard Error of Mean 0.011

4. Secondary Outcome: FEV1 AUC0-6 at Day 1
Description: Area between the test-day baseline FEV1 and the FEV1 change from the test-day baseline curve from 0 to 6 hours divided by 6 at Day 1
Time Frame: Before drug administration to 6 hours after drug administration on Day 1
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.173 (0.008) | 0.189 (0.008) | 0.124 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established for this comparison; p = 0.124, ANCOVA; Mean Difference (Final Values) = -0.016, 95% CI [-0.036 to 0.004], Standard Error of Mean 0.010

5. Secondary Outcome: FEV1 AUC0-6 at Day 29
Description: Area between the test-day baseline FEV1 and the FEV1 change from the test-day baseline curve from 0 to 6 hours divided by 6 at Day 29
Time Frame: Before drug administration to 6 hours after drug administration on Day 29
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.154 (0.007) | 0.161 (0.007) | 0.127 (0.007)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established for this comparison; p = 0.4888, ANCOVA; Mean Difference (Final Values) = -0.007, 95% CI [-0.026 to 0.013], Standard Error of Mean 0.01

6. Secondary Outcome: FEV1 AUC0-6 at Day 57
Description: Area between the test-day baseline FEV1 and the FEV1 change from the test-day baseline curve from 0 to 6 hours divided by 6 at Day 57
Time Frame: Before drug administration to 6 hours after drug administration on Day 57
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.146 (0.007) | 0.16 (0.007) | 0.118 (0.007)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established for this comparison; p = 0.1433, ANCOVA; Mean Difference (Final Values) = -0.014, 95% CI [-0.033 to 0.005]

7. Secondary Outcome: FEV1 AUC0-4 at Day 1
Description: Area between the test-day baseline FEV1 and the FEV1 change from the test-day baseline curve from 0 to 4 hours divided by 4 at Day 1
Time Frame: Before drug administration to 4 hours after drug administration on Day 1
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.211 (0.008) | 0.227 (0.008) | 0.149 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.061, 95% CI [0.04 to 0.083], Standard Error of Mean 0.011

8. Secondary Outcome: FEV1 AUC0-4 at Day 29
Description: Area between the test-day baseline FEV1 and the FEV1 change from the test-day baseline curve from 0 to 4 hours divided by 4 at Day 29
Time Frame: Before drug administration to 4 hours after drug administration on Day 29
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.197 (0.008) | 0.198 (0.008) | 0.153 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.044, 95% CI [0.024 to 0.065], Standard Error of Mean 0.01

9. Secondary Outcome: FEV1 AUC0-4 at Day 57
Description: Area between the test-day baseline FEV1 and the FEV1 change from the test-day baseline curve from 0 to 4 hours divided by 4 at Day 57
Time Frame: Before drug administration to 4 hours after drug administration on Day 57
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.188 (0.007) | 0.200 (0.007) | 0.141 (0.007)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.047, 95% CI [0.027 to 0.067], Standard Error of Mean 0.01

10. Secondary Outcome: FEV1 AUC4-6 at Day 1
Description: Area between the test-day baseline FEV1 and the FEV1 change from the test-day baseline curve from 4 to 6 hours divided by 2 at Day 1
Time Frame: Between 4 hours and 6 hours after drug administration on Day 1
Population: Full Analysis Set for Pulmonary Function Test Data 4-6 hours
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 447 | 449 | 427
liters | 0.1 (0.008) | 0.115 (0.009) | 0.074 (0.009)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.0258, ANCOVA; Mean Difference (Final Values) = 0.026, 95% CI [0.003 to 0.049], Standard Error of Mean 0.012

11. Secondary Outcome: FEV1 AUC4-6 at Day 29
Description: Area between the test-day baseline FEV1 and the FEV1 change from the test-day baseline curve from 4 to 6 hours divided by 2 at Day 29
Time Frame: Between 4 hours and 6 hours after drug administration on Day 29
Population: Full Analysis Set for Pulmonary Function Test Data 4-6 hours
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 447 | 449 | 427
liters | 0.068 (0.008) | 0.087 (0.008) | 0.078 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.3749, ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI [-0.032 to 0.012], Standard Error of Mean 0.011

12. Secondary Outcome: FEV1 AUC4-6 at Day 57
Description: Area between the test-day baseline FEV1 and the FEV1 change from the test-day baseline curve from 4 to 6 hours divided by 2 at Day 57
Time Frame: Between 4 hours and 6 hours after drug administration on Day 57
Population: Full Analysis Set for Pulmonary Function Test Data 4-6 hours
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 447 | 449 | 427
liters | 0.063 (0.008) | 0.084 (0.008) | 0.073 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.3355, ANCOVA; Mean Difference (Final Values) = -0.011, 95% CI [-0.033 to 0.011], Standard Error of Mean 0.011

13. Secondary Outcome: Peak FEV1 Response at Day 1
Description: Maximum change in recorded FEV1 value from the corresponding test-day baseline within the first 2 hours after drug administration on Day 1
Time Frame: Within the first 2-hour post-treatment interval on Day 1
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.302 (0.008) | 0.323 (0.008) | 0.237 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.0743, ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI [-0.042 to 0.002], Standard Error of Mean 0.011

14. Secondary Outcome: Peak FEV1 Response at Day 29
Description: Maximum change in recorded FEV1 value from the corresponding test-day baseline within the first 2 hours after drug administration on Day 29
Time Frame: Within the first 2-hour post-treatment interval on Day 29
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.302 (0.008) | 0.296 (0.008) | 0.237 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.5711, ANCOVA; Mean Difference (Final Values) = 0.006, 95% CI [-0.015 to 0.028], Standard Error of Mean 0.011

15. Secondary Outcome: Peak FEV1 Response at Day 57
Description: Maximum change in recorded FEV1 value from the corresponding test-day baseline within the first 2 hours after drug administration on Day 57
Time Frame: Within the first 2-hour post-treatment interval on Day 57
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.284 (0.008) | 0.296 (0.008) | 0.223 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.2274, ANCOVA; Mean Difference (Final Values) = -0.013, 95% CI [-0.033 to 0.008], Standard Error of Mean 0.011

16. Secondary Outcome: Peak FEV1 Response at Day 85
Description: Maximum change in recorded FEV1 value from the corresponding test-day baseline within the first 2 hours after drug administration on Day 85
Time Frame: Within the first 2-hour post-treatment interval on Day 85
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.293 (0.008) | 0.290 (0.008) | 0.225 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.8065, ANCOVA; Mean Difference (Final Values) = 0.003, 95% CI [-0.018 to 0.024], Standard Error of Mean 0.011

17. Secondary Outcome: Peak FEV1 Response at Day 1
Description: as for outcome 13
Time Frame: Within the first 2-hour post-treatment interval on Day 1
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.302 (0.008) | 0.323 (0.008) | 0.237 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.065, 95% CI [0.043 to 0.087], Standard Error of Mean 0.011

18. Secondary Outcome: Peak FEV1 Response at Day 29
Description: as for outcome 14
Time Frame: Within the first 2-hour post-treatment interval on Day 29
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.302 (0.008) | 0.296 (0.008) | 0.237 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.065, 95% CI [0.044 to 0.087], Standard Error of Mean 0.011

19. Secondary Outcome: Peak FEV1 Response at Day 57
Description: as for outcome 15
Time Frame: Within the first 2-hour post-treatment interval on Day 57
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.284 (0.008) | 0.296 (0.008) | 0.223 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.06, 95% CI [0.04 to 0.081], Standard Error of Mean 0.011

20. Secondary Outcome: Peak FEV1 Response at Day 85
Description: as for outcome 16
Time Frame: Within the first 2-hour post-treatment interval on Day 85
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.293 (0.008) | 0.290 (0.008) | 0.225 (0.008)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.068, 95% CI [0.047 to 0.089], Standard Error of Mean 0.011

21. Secondary Outcome: Time to Onset of Therapeutic FEV1 Response at Day 1
Description: Achievement of recorded FEV1 measurement of at least 1.15 times of the corresponding test-day baseline value at any time during the first 2 hours of observation after drug administration at Day 1
Time Frame: Within the first 2-hour post-treatment interval at Day 1
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
Minutes | 13 (NA) [8 to 59] | 12 (NA) [7 to 48] | 28 (NA) [11 to 361]

22. Secondary Outcome: Time to Onset of Therapeutic FEV1 Response at Day 29
Description: Achievement of recorded FEV1 measurement of at least 1.15 times of the corresponding test-day baseline value at any time during the first 2 hours of observation after drug administration at Day 29
Time Frame: Within the first 2-hour post-treatment interval at Day 29
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
Minutes | 12 (NA) [7 to 53] | 13 (NA) [8 to 55] | 27 (NA) [11 to 361]

23. Secondary Outcome: Time to Onset of Therapeutic FEV1 Response at Day 57
Description: Achievement of recorded FEV1 measurement of at least 1.15 times of the corresponding test-day baseline value at any time during the first 2 hours of observation after drug administration at Day 57
Time Frame: Within the first 2-hour post-treatment interval at Day 57
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
Minutes | 13 (NA) [8 to 361] | 12 (NA) [7 to 59] | 29 (NA) [11 to 361]

24. Secondary Outcome: Time to Onset of Therapeutic FEV1 Response at Day 85
Description: Achievement of recorded FEV1 measurement of at least 1.15 times of the corresponding test-day baseline value at any time during the first 2 hours of observation after drug administration at Day 85
Time Frame: Within the first 2-hour post-treatment interval at Day 85
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
Minutes | 12 (NA) [8 to 102] | 13 (NA) [8 to 361] | 27 (NA) [11 to 361]

25. Secondary Outcome: Duration of Therapeutic FEV1 Response at Day 1
Description: The time interval between the onset and the the termination of a therapeutic FEV1 response (at least 1.15 times the corresponding test-day baseline value) during the 6-hour observation period at Day 1
Time Frame: During the 6-hour observation period after drug administration at Day 1
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
Minutes | 189 (NA) [29 to 323] | 219 (NA) [42 to 336] | 104 (NA) [0 to 309]

26. Secondary Outcome: Duration of Therapeutic FEV1 Response at Day 29
Description: The time interval between the onset and the the termination of a therapeutic FEV1 response (at least 1.15 times the corresponding test-day baseline value) during the 6-hour observation period at Day 29
Time Frame: During the 6-hour observation period after drug administration at Day 29
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
Minutes | 170 (NA) [16 to 298] | 178 (NA) [11 to 306] | 122 (NA) [0 to 312]

27. Secondary Outcome: Duration of Therapeutic FEV1 Response at Day 57
Description: The time interval between the onset and the the termination of a therapeutic FEV1 response (at least 1.15 times the corresponding test-day baseline value) during the 6-hour observation period at Day 57
Time Frame: During the 6-hour observation period after drug administration at Day 57
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
Minutes | 165 (NA) [0 to 288] | 194 (NA) [11 to 318] | 84 (NA) [0 to 303]

28. Secondary Outcome: Duration of Therapeutic FEV1 Response at Day 85
Description: The time interval between the onset and the the termination of a therapeutic FEV1 response (at least 1.15 times the corresponding test-day baseline value) during the 6-hour observation period at Day 85
Time Frame: During the 6-hour observation period after drug administration at Day 85
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
Minutes | 168 (NA) [1 to 284] | 172 (NA) [0 to 302] | 70 (NA) [0 to 285]

29. Secondary Outcome: Time to Peak FEV1 Response at Day 1
Description: The first time point at which the maximum change in recorded FEV1 data from the corresponding test-day baseline occurred during the 6-hours observation period after drug administration at Day 1
Time Frame: Within the 6-hour post-treatment observation period at Day 1
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
Minutes | 60 (NA) [30 to 120] | 60 (NA) [60 to 120] | 120 (NA) [60 to 180]

30. Secondary Outcome: Time to Peak FEV1 Response at Day 29
Description: The first time point at which the maximum change in recorded FEV1 data from the corresponding test-day baseline occurred during the 6-hours observation period after drug administration at Day 29
Time Frame: Within the 6-hour post-treatment observation period at Day 29
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
Minutes | 60 (NA) [30 to 120] | 60 (NA) [30 to 120] | 120 (NA) [45 to 180]

31. Secondary Outcome: Time to Peak FEV1 Response at Day 57
Description: The first time point at which the maximum change in recorded FEV1 data from the corresponding test-day baseline occurred during the 6-hours observation period after drug administration at Day 57
Time Frame: Within the 6-hour post-treatment observation period at Day 57
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
Minutes | 60 (NA) [30 to 120] | 60 (NA) [30 to 120] | 60 (NA) [30 to 180]

32. Secondary Outcome: Time to Peak FEV1 Response at Day 85
Description: The first time point at which the maximum change in recorded FEV1 data from the corresponding test-day baseline occurred during the 6-hours observation period after drug administration at Day 85
Time Frame: Within the 6-hour post-treatment observation period at Day 85
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
Minutes | 60 (NA) [30 to 120] | 60 (NA) [30 to 120] | 60 (NA) [30 to 180]

33. Secondary Outcome: FVC AUC0-6 at Day 1
Description: Area between the test-day baseline FVC and the FVC change from the test-day baseline curve from 0 to 6 hours divided by 6 at Day 1
Time Frame: Before drug administration to 6 hours after drug administration at Day 1
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.337 (0.015) | 0.354 (0.015) | 0.25 (0.016)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.417, ANCOVA; Mean Difference (Final Values) = -0.017, 95% CI [-0.058 to 0.024], Standard Error of Mean 0.021

34. Secondary Outcome: FVC AUC0-6 at Day 29
Description: Area between the test-day baseline FVC and the FVC change from the test-day baseline curve from 0 to 6 hours divided by 6 at Day 29
Time Frame: Before drug administration to 6 hours after drug administration at Day 29
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.3 (0.015) | 0.319 (0.015) | 0.246 (0.015)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.3505, ANCOVA; Mean Difference (Final Values) = -0.019, 95% CI [-0.059 to 0.021], Standard Error of Mean 0.02

35. Secondary Outcome: FVC AUC0-6 at Day 57
Description: Area between the test-day baseline FVC and the FVC change from the test-day baseline curve from 0 to 6 hours divided by 6 at Day 57
Time Frame: Before drug administration to 6 hours after drug administration on Day 57
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.284 (0.015) | 0.303 (0.015) | 0.22 (0.015)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.3499, ANCOVA; Mean Difference (Final Values) = -0.019, 95% CI [-0.058 to 0.021], Standard Error of Mean 0.02

36. Secondary Outcome: FVC AUC0-6 at Day 85
Description: Area between the test-day baseline FVC and the FVC change from the test-day baseline curve from 0 to 6 hours divided by 6 at Day 85
Time Frame: Before drug administration to 6 hours after drug administration on Day 85
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.279 (0.015) | 0.283 (0.015) | 0.219 (0.015)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.8288, ANCOVA; Mean Difference (Final Values) = -0.004, 95% CI [-0.044 to 0.035], Standard Error of Mean 0.02

37. Secondary Outcome: FVC AUC0-4 at Day 1
Description: Area between the test-day baseline FVC and the FVC change from the test-day baseline curve from 0 to 4 hours divided by 4 at Day 1
Time Frame: Before drug administration to 4 hours after drug administration on Day 1
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.408 (0.016) | 0.422 (0.016) | 0.297 (0.016)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.112, 95% CI [0.069 to 0.154], Standard Error of Mean 0.022

38. Secondary Outcome: FVC AUC0-4 at Day 29
Description: Area between the test-day baseline FVC and the FVC change from the test-day baseline curve from 0 to 4 hours divided by 4 at Day 29
Time Frame: Before drug administration to 4 hours after drug administration on Day 29
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.381 (0.015) | 0.388 (0.015) | 0.291 (0.016)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.09, 95% CI [0.049 to 0.132], Standard Error of Mean 0.021

39. Secondary Outcome: FVC AUC0-4 at Day 57
Description: Area between the test-day baseline FVC and the FVC change from the test-day baseline curve from 0 to 4 hours divided by 4 at Day 57
Time Frame: Before drug administration to 4 hours after drug administration on Day 57
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.361 (0.015) | 0.380 (0.015) | 0.264 (0.015)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.097, 95% CI [0.056 to 0.138], Standard Error of Mean 0.021

40. Secondary Outcome: FVC AUC0-4 at Day 85
Description: Area between the test-day baseline FVC and the FVC change from the test-day baseline curve from 0 to 4 hours divided by 4 at Day 85
Time Frame: Before drug administration to 4 hours after drug administration on Day 85
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.359 (0.015) | 0.359 (0.015) | 0.265 (0.015)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.094, 95% CI [0.054 to 0.135], Standard Error of Mean 0.021

41. Secondary Outcome: FVC AUC4-6 at Day 1
Description: Area between the test-day baseline FVC and the FVC change from the test-day baseline curve from 4 to 6 hours divided by 2 at Day 1
Time Frame: Between 4 hours and 6 hours after drug administration on Day 1
Population: Full Analysis Set for Pulmonary Function Test Data 4-6 hours
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 447 | 449 | 427
liters | 0.2 (0.017) | 0.221 (0.017) | 0.156 (0.018)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.0688, ANCOVA; Mean Difference (Final Values) = 0.043, 95% CI [-0.003 to 0.09], Standard Error of Mean 0.024

42. Secondary Outcome: FVC AUC4-6 at Day 29
Description: Area between the test-day baseline FVC and the FVC change from the test-day baseline curve from 4 to 6 hours divided by 2 at Day 29
Time Frame: Between 4 hours and 6 hours after drug administration on Day 29
Population: Full Analysis Set for Pulmonary Function Test Data 4-6 hours
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 447 | 449 | 427
liters | 0.137 (0.017) | 0.180 (0.017) | 0.156 (0.017)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.3895, ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI [-0.064 to 0.025], Standard Error of Mean 0.023

43. Secondary Outcome: FVC AUC4-6 at Day 57
Description: Area between the test-day baseline FVC and the FVC change from the test-day baseline curve from 4 to 6 hours divided by 2 at Day 57
Time Frame: Between 4 hours and 6 hours after drug administration on Day 57
Population: Full Analysis Set for Pulmonary Function Test Data 4-6 hours
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 447 | 449 | 427
liters | 0.128 (0.016) | 0.147 (0.016) | 0.13 (0.017)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.959, ANCOVA; Mean Difference (Final Values) = -0.001, 95% CI [-0.045 to 0.042], Standard Error of Mean 0.022

44. Secondary Outcome: FVC AUC4-6 at Day 85
Description: Area between the test-day baseline FVC and the FVC change from the test-day baseline curve from 4 to 6 hours divided by 2 at Day 85
Time Frame: Between 4 hours and 6 hours after drug administration on Day 85
Population: Full Analysis Set for Pulmonary Function Test Data 4-6 hours
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 447 | 449 | 427
liters | 0.117 (0.017) | 0.130 (0.017) | 0.124 (0.017)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.7652, ANCOVA; Mean Difference (Final Values) = -0.007, 95% CI [-0.053 to 0.039], Standard Error of Mean 0.023

45. Secondary Outcome: Peak FVC Response at Day 1
Description: Maximum change in recorded FVC value from the corresponding test-day baseline within the first 2 hours after drug administration on Day 1
Time Frame: Within the first 2-hour post-treatment interval at Day 1
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.6 (0.017) | 0.612 (0.017) | 0.479 (0.017)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.6244, ANCOVA; Mean Difference (Final Values) = -0.011, 95% CI [-0.057 to 0.034], Standard Error of Mean 0.023

46. Secondary Outcome: Peak FVC Response at Day 29
Description: Maximum change in recorded FVC value from the corresponding test-day baseline within the first 2 hours after drug administration on Day 29
Time Frame: Within the first 2-hour post-treatment interval at Day 29
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.594 (0.017) | 0.591 (0.017) | 0.465 (0.017)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.873, ANCOVA; Mean Difference (Final Values) = 0.004, 95% CI [-0.041 to 0.049], Standard Error of Mean 0.023

47. Secondary Outcome: Peak FVC Response at Day 57
Description: Maximum change in recorded FVC value from the corresponding test-day baseline within the first 2 hours after drug administration on Day 57
Time Frame: Within the first 2-hour post-treatment interval at Day 57
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.562 (0.017) | 0.577 (0.017) | 0.445 (0.017)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.5294, ANCOVA; Mean Difference (Final Values) = -0.015, 95% CI [-0.06 to 0.031], Standard Error of Mean 0.023

48. Secondary Outcome: Peak FVC Response at Day 85
Description: Maximum change in recorded FVC value from the corresponding test-day baseline within the first 2 hours after drug administration on Day 85
Time Frame: Within the first 2-hour post-treatment interval at Day 85
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.575 (0.017) | 0.562 (0.017) | 0.449 (0.017)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.563, ANCOVA; Mean Difference (Final Values) = 0.013, 95% CI [-0.032 to 0.058], Standard Error of Mean 0.023

49. Secondary Outcome: Peak FVC Response at Day 1
Description: as for outcome 45
Time Frame: Within the first 2-hour post-treatment interval at Day 1
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.6 (0.017) | 0.612 (0.017) | 0.479 (0.017)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.121, 95% CI [0.075 to 0.167], Standard Error of Mean 0.024

50. Secondary Outcome: Peak FVC Response at Day 29
Description: as for outcome 46
Time Frame: Within the first 2-hour post-treatment interval at Day 29
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.594 (0.017) | 0.591 (0.017) | 0.465 (0.017)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.129, 95% CI [0.084 to 0.174], Standard Error of Mean 0.023

51. Secondary Outcome: Peak FVC Response at Day 57
Description: as for outcome 47
Time Frame: Within the first 2-hour post-treatment interval at Day 57
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.562 (0.017) | 0.577 (0.017) | 0.445 (0.017)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.118, 95% CI [0.072 to 0.163], Standard Error of Mean 0.023

52. Secondary Outcome: Peak FVC Response at Day 85
Description: as for outcome 48
Time Frame: Within the first 2-hour post-treatment interval at Day 85
Population: Full Analysis Set for Pulmonary Function Test Data
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 474 | 482 | 468
liters | 0.575 (0.017) | 0.562 (0.017) | 0.449 (0.017)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = 0.126, 95% CI [0.081 to 0.171], Standard Error of Mean 0.023

53. Secondary Outcome: Rescue Medication Use on Pulmonary Test Day 1
Description: Number of patients used rescue medication during the 6-hour pulmonary function testing after drug administration on Day 1
Time Frame: During the 6-hour pulmonary function testing after drug administration on Day 1
Population: Treated Set
Measure: Number; unit: patients
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 486 | 491 | 483
patients | 8 | 9 | 7

54. Secondary Outcome: Rescue Medication Use on Pulmonary Test Day 29
Description: Number of patients used rescue medication during the 6-hour pulmonary function testing after drug administration on Day 29
Time Frame: During the 6-hour pulmonary function testing after drug administration on Day 29
Population: Treated Set
Measure: Number; unit: patients
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 486 | 491 | 483
patients | 10 | 7 | 7

55. Secondary Outcome: Rescue Medication Use on Pulmonary Test Day 57
Description: Number of patients used rescue medication during the 6-hour pulmonary function testing after drug administration on Day 57
Time Frame: During the 6-hour pulmonary function testing after drug administration on Day 57
Population: Treated Set
Measure: Number; unit: patients
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 486 | 491 | 483
patients | 7 | 7 | 6

56. Secondary Outcome: Rescue Medication Use on Pulmonary Test Day 85
Description: Number of patients used rescue medication during the 6-hour pulmonary function testing after drug administration on Day 85
Time Frame: During the 6-hour pulmonary function testing after drug administration on Day 85
Population: Treated Set
Measure: Number; unit: patients
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 486 | 491 | 483
patients | 5 | 7 | 10

57. Secondary Outcome: Night-time Rescue Medication Use
Description: The mean number of puffs of rescue medication used during the night-time per week during the entire study (including baseline and on-treatment period)
Time Frame: During the 2-week baseline washout period and the 12-week treatment period
Population: Full Analysis Set for Diary Data
Measure: Least Squares Mean (Standard Error); unit: puffs
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 471 | 467 | 454
puffs | 0.977 (0.047) | 0.977 (0.047) | 0.997 (0.048)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.9943, ANCOVA; Mean Difference (Final Values) = -0.00045, 95% CI [-0.1259 to 0.125], Standard Error of Mean 0.06396
Statistical Analysis 2: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p = 0.7569, ANCOVA; Mean Difference (Final Values) = -0.01995, 95% CI 2-sided [-0.1463 to 0.1064], Standard Error of Mean 0.06441

58. Secondary Outcome: Daytime Rescue Medication Use
Description: The mean number of puffs of rescue medication used during the daytime per week during the entire study (including baseline and on-treatment period)
Time Frame: During the 2-week baseline washout period and the 12-week treatment period
Population: Full Analysis Set for Diary Data
Measure: Least Squares Mean (Standard Error); unit: puffs
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 453 | 458 | 438
puffs | 2.3 (0.089) | 2.191 (0.089) | 2.456 (0.09)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.3659, ANCOVA; Mean Difference (Final Values) = 0.1091, 95% CI [-0.1276 to 0.3458], Standard Error of Mean 0.1206
Statistical Analysis 2: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p = 0.203, ANCOVA; Mean Difference (Final Values) = -0.1554, 95% CI 2-sided [-0.3947 to 0.08395], Standard Error of Mean 0.122

59. Secondary Outcome: Night-time Symptom Score
Description: The weekly mean night-time symptom score per week during the entire study (including baseline and on-treatment period).
  Night-time COPD symptoms: 0=none 1=some - slept well 2=woke once 3=woke several times 4=woke most of night
Time Frame: During the 2-week baseline washout period and the 12-week treatment period
Population: Full Analysis Set for Diary Data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 471 | 467 | 454
units on a scale | 0.922 (0.023) | 0.914 (0.024) | 0.857 (0.024)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.809, ANCOVA; Mean Difference (Final Values) = 0.007734, 95% CI [-0.05503 to 0.0705], Standard Error of Mean 0.03199
Statistical Analysis 2: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p = 0.044, ANCOVA; Mean Difference (Final Values) = 0.06501, 95% CI 2-sided [0.001746 to 0.1283], Standard Error of Mean 0.03225

60. Secondary Outcome: Daytime Symptom Score
Description: The weekly mean daytime symptom score per week during the entire study (including baseline and on-treatment period).
  Daytime COPD symptoms: 0=none 1=occasional 2=frequent, no interference with activities 3=most of day, interference with activities 4=prevent working and activities
Time Frame: During the 2-week baseline washout period and the 12-week treatment period
Population: Full Analysis Set for Diary Data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 452 | 456 | 437
units on a scale | 1.015 (0.022) | 1.002 (0.022) | 0.999 (0.022)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.6674, ANCOVA; Mean Difference (Final Values) = 0.0129, 95% CI [-0.04598 to 0.07179], Standard Error of Mean 0.03002
Statistical Analysis 2: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p = 0.604, ANCOVA; Mean Difference (Final Values) = 0.01573, 95% CI 2-sided [-0.04376 to 0.07523], Standard Error of Mean 0.03033

61. Secondary Outcome: Trough Peak Expiratory Flow Rate (PEFR)
Description: The weekly mean trough PEFR during the entire study (including baseline and on-treatment period)
Time Frame: During the 2-week baseline washout period and the 12-week treatment period and PEFR taken before administration of study medication
Population: Full Analysis Set for Diary Data
Measure: Least Squares Mean (Standard Error); unit: liters/min
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 441 | 444 | 426
liters/min | 191.95 (1.51) | 190.290 (1.526) | 189.51 (1.551)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.4238, ANCOVA; Mean Difference (Final Values) = 1.6526, 95% CI [-2.3995 to 5.7047], Standard Error of Mean 2.0653
Statistical Analysis 2: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p = 0.2431, ANCOVA; Mean Difference (Final Values) = 2.4376, 95% CI 2-sided [-1.6578 to 6.533], Standard Error of Mean 2.0874

62. Secondary Outcome: Physician's Global Evaluation Score on Pulmonary Function Testing Day 29
Description: Physician's Global Evaluation score is based on the need for concomitant medication, number and severity of exacerbations since the last visit, severity of cough, ability to exercise, amount of wheezing, etc.
  Score: 1,2 = poor; 3,4 = fair; 5,6 =good; 7,8 = excellent.
Time Frame: Prior to pulmonary function test on Day 29
Population: Treated Set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 480 | 487 | 481
units on a scale | 4.936 (0.041) | 4.859 (0.041) | 4.99 (0.041)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.173, ANCOVA; Mean Difference (Final Values) = 0.077, 95% CI [-0.034 to 0.187], Standard Error of Mean 0.056
Statistical Analysis 2: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p = 0.336, ANCOVA; Mean Difference (Final Values) = -0.054, 95% CI 2-sided [-0.165 to 0.056], Standard Error of Mean 0.056

63. Secondary Outcome: Physician's Global Evaluation Score on Pulmonary Function Testing Day 57
Description: as for outcome 62
Time Frame: Prior to pulmonary function test on Day 57
Population: Treated Set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 480 | 487 | 481
units on a scale | 4.971 (0.045) | 4.965 (0.045) | 5.04 (0.046)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.924, ANCOVA; Mean Difference (Final Values) = 0.006, 95% CI [-0.115 to 0.127], Standard Error of Mean 0.062
Statistical Analysis 2: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p = 0.266, ANCOVA; Mean Difference (Final Values) = -0.069, 95% CI 2-sided [-0.19 to 0.053], Standard Error of Mean 0.062

64. Secondary Outcome: Physician's Global Evaluation Score on Pulmonary Function Testing Day 85
Description: as for outcome 62
Time Frame: Prior to pulmonary function test on Day 85
Population: Treated Set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 480 | 487 | 481
units on a scale | 5.115 (0.048) | 5.018 (0.048) | 5.097 (0.048)
Statistical Analysis 1: Comparison: COMBIVENT Respimat 20/100 mcg vs COMBIVENT CFC-MDI 36/206 mcg; Test type: Non-Inferiority or Equivalence — This analysis is purely exploratory. Non-inferiority margin is not established; p = 0.139, ANCOVA; Mean Difference (Final Values) = 0.097, 95% CI [-0.031 to 0.225], Standard Error of Mean 0.065
Statistical Analysis 2: Comparison: COMBIVENT Respimat 20/100 mcg vs Ipratropium Respimat 20 mcg; This analysis is purely exploratory; Test type: Superiority or Other; p = 0.788, ANCOVA; Mean Difference (Final Values) = 0.018, 95% CI 2-sided [-0.111 to 0.146], Standard Error of Mean 0.066

65. Secondary Outcome: Percentage of Patients With Chronic Obstructive Pulmonary Disease (COPD) Exacerbation During the On-treatment Period
Description: COPD exacerbation is defined as an increase or new onset of more than one of the following respiratory symptoms (cough, sputum, sputum purulence, wheezing, dyspnea, and chest tightness) having a duration of three or more days requiring treatment with an antibiotic and/or systemic steroids with or without hospital admission.
Time Frame: During the 12-week on-treatment period
Population: Treated Set
Measure: Number; unit: Percentage of patients
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 486 | 491 | 483
Percentage of patients | 14.81 | 13.03 | 10.35

66. Secondary Outcome: COPD Exacerbation Rate During the On-treatment Period
Description: Proportion of patients experiencing a COPD exacerbation per patient year. COPD exacerbation is defined as an increase or new onset of more than one of the following respiratory symptoms (cough, sputum, sputum purulence, wheezing, dyspnea, and chest tightness) having a duration of three or more days requiring treatment with an antibiotic and/or systemic steroids with or without hospital admission.
Time Frame: During the 12-week on-treatment period
Population: Treated Set
Measure: Number; unit: Proportion of patients
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 486 | 491 | 483
Proportion of patients | 0.76 (NA) | 0.69 (NA) | 0.53 (NA)

67. Secondary Outcome: COPD Exacerbation During the On-treatment Period
Description: as for outcome 65
Time Frame: During the 12-week on-treatment period
Population: Treated Set
Measure: Number; unit: Percentage of patients
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 486 | 491 | 483
Percentage of patients | 3.27 | 2.93 | 2.13

68. Secondary Outcome: Frequency Distribution of Satisfaction Rating With Inhaler Attributes
Time Frame: 12 weeks
Population: Treated set (US patients)
Measure: Number; unit: participants
Groups:
- MDI Device: MDI Inhalers
- RESPIMAT Device: Respimat Inhalers
Arm/Group | MDI Device | RESPIMAT Device
Number analyzed (Participants) | 834 | 835
participants
  Very dissatisfied | 16 | 13
  Dissatisfied | 27 | 20
  Somewhat dissatisfied | 37 | 17
  Satisfied/dissatisfied | 54 | 27
  Somewhat satisfied | 109 | 46
  Satisfied | 351 | 305
  Very satisfied | 240 | 407

69. Secondary Outcome: Mean Rating Scores of Satisfaction With Inhaler - Overall Feeling of Inhaling Medicine
Description: Patients rated their response on a seven point Likert scale:
  1 = very dissatisfied, 2 = dissatisfied, 3 = somewhat dissatisfied, 4 = neither satisfied nor dissatisfied, 5 = somewhat satisfied, 6 = satisfied, 7 = very satisfied.
Time Frame: 12 weeks
Population: Treated set (US patients)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MDI Device | RESPIMAT Device
Number analyzed (Participants) | 834 | 835
units on a scale | 5.411 (0.049) | 5.810 (0.049)
Statistical Analysis 1: Comparison: MDI Device vs RESPIMAT Device; Difference: Respimat - MDI; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.398, Standard Error of Mean 0.065

70. Secondary Outcome: Mean Rating Scores of Satisfaction With Inhaler - Feeling That the Inhaled Dose Goes to the Lung
Description: as for outcome 69
Time Frame: 12 weeks
Population: Treated set (US patients)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MDI Device | RESPIMAT Device
Number analyzed (Participants) | 833 | 835
units on a scale | 5.326 (0.049) | 5.808 (0.049)
Statistical Analysis 1: Comparison: MDI Device vs RESPIMAT Device; Difference: Respimat - MDI; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.482, Standard Error of Mean 0.065

71. Secondary Outcome: Mean Rating Scores of Satisfaction With Inhaler - Telling the Amount of Medication Left
Description: as for outcome 69
Time Frame: 12 weeks
Population: Treated set (US patients)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MDI Device | RESPIMAT Device
Number analyzed (Participants) | 833 | 835
units on a scale | 4.573 (0.057) | 6.184 (0.057)
Statistical Analysis 1: Comparison: MDI Device vs RESPIMAT Device; Difference: Respimat - MDI; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 1.612, Standard Error of Mean 0.075

72. Secondary Outcome: Mean Rating Scores of Satisfaction With Inhaler - The Inhaler Works Reliably
Description: as for outcome 69
Time Frame: 12 weeks
Population: Treated set (US patients)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MDI Device | RESPIMAT Device
Number analyzed (Participants) | 834 | 835
units on a scale | 5.682 (0.044) | 6.190 (0.044)
Statistical Analysis 1: Comparison: MDI Device vs RESPIMAT Device; Difference: Respimat - MDI; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.508, Standard Error of Mean 0.058

73. Secondary Outcome: Mean Rating Scores of Satisfaction With Inhaler - Ease of Inhaling a Dose From the Inhaler
Description: as for outcome 69
Time Frame: 12 weeks
Population: Treated set (US patients)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MDI Device | RESPIMAT Device
Number analyzed (Participants) | 834 | 835
units on a scale | 5.729 (0.046) | 6.150 (0.046)
Statistical Analysis 1: Comparison: MDI Device vs RESPIMAT Device; Difference: Respimat - MDI; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.421, Standard Error of Mean 0.061

74. Secondary Outcome: Mean Rating Scores of Satisfaction With Inhaler - Instructions for Use
Description: as for outcome 69
Time Frame: 12 weeks
Population: Treated set (US patients)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MDI Device | RESPIMAT Device
Number analyzed (Participants) | 834 | 834
units on a scale | 6.048 (0.036) | 6.275 (0.036)
Statistical Analysis 1: Comparison: MDI Device vs RESPIMAT Device; Difference: Respimat - MDI; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.226, Standard Error of Mean 0.047

75. Secondary Outcome: Mean Rating Scores of Satisfaction With Inhaler - The Inhaler is Durable
Description: as for outcome 69
Time Frame: 12 weeks
Population: Treated set (US patients)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MDI Device | RESPIMAT Device
Number analyzed (Participants) | 834 | 835
units on a scale | 6.014 (0.037) | 6.279 (0.037)
Statistical Analysis 1: Comparison: MDI Device vs RESPIMAT Device; Difference: Respimat - MDI; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.265, Standard Error of Mean 0.050

76. Secondary Outcome: Mean Rating Scores of Satisfaction With Inhaler - Using the Inhaler
Description: as for outcome 69
Time Frame: 12 weeks
Population: Treated set (US patients)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MDI Device | RESPIMAT Device
Number analyzed (Participants) | 833 | 835
units on a scale | 5.749 (0.045) | 6.127 (0.045)
Statistical Analysis 1: Comparison: MDI Device vs RESPIMAT Device; Difference: Respimat - MDI; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.378, Standard Error of Mean 0.060

77. Secondary Outcome: Mean Rating Scores of Satisfaction With Inhaler - Speed of Medicine Coming Out of the Inhaler
Description: as for outcome 69
Time Frame: 12 weeks
Population: Treated set (US patients)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MDI Device | RESPIMAT Device
Number analyzed (Participants) | 834 | 835
units on a scale | 5.715 (0.047) | 6.117 (0.047)
Statistical Analysis 1: Comparison: MDI Device vs RESPIMAT Device; Difference: Respimat - MDI; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.402, Standard Error of Mean 0.062

78. Secondary Outcome: Mean Rating Scores of Satisfaction With Inhaler - Overall Satisfaction With Inhaler
Description: as for outcome 69
Time Frame: 12 weeks
Population: Treated set (US patients)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | MDI Device | RESPIMAT Device
Number analyzed (Participants) | 834 | 835
units on a scale | 5.639 (0.048) | 6.103 (0.048)
Statistical Analysis 1: Comparison: MDI Device vs RESPIMAT Device; Difference: Respimat - MDI; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = 0.464, Standard Error of Mean 0.063

79. Secondary Outcome: Device Preference (Respimat or MDI)
Description: Frequency of patients due to device preference
Time Frame: 12 weeks
Population: Treated set (US patients)
Measure: Number; unit: participants
Groups:
- Number of Patients: Total number of patients due to device preference
Arm/Group | Number of Patients
Number analyzed (Participants) | 835
participants
  Prefer Respimat | 584
  Prefer MDI | 146
  No preference | 105

80. Secondary Outcome: Rating of Action of Turning Clear Base of Respimat
Description: Frequency of patients due to rating of action of turning clear base of Respimat
Time Frame: 12 weeks
Population: Treated set (US patients)
Measure: Number; unit: participants
Groups:
- Number of Patients: Total number of patients due to rating of turning
Arm/Group | Number of Patients
Number analyzed (Participants) | 835
participants
  Very easy | 587
  Easy | 204
  Neither easy nor difficult | 40
  Difficult | 4
  Very difficult | 0

81. Secondary Outcome: Noncompartmental Pharmacokinetic Parameters of Ipratropium at Steady State
Description: Geometric mean area under the plasma drug concentration time curve over one dosing interval (AUCτ). Each patient had eight plasma samples (trough pre-dose, 5, 15, 30, and 60 minutes post-dose, as well as 2, 4, and 6 hours post-dose).
Time Frame: Before drug administration to 6 hours after drug administration on Day 29
Population: All patients in FAS who were from U.S. study sites and whose blood and/or urine samples were collected at Visit 3 according to the protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 43 | 49 | 48
pg*h/mL | 128 (55.4) | 123 (79.3) | 115 (50.9)

82. Secondary Outcome: Noncompartmental Parameters of Albuterol at Steady State
Description: as for outcome 81
Time Frame: Before drug administration to 6 hours after drug administration on Day 29
Population: as for outcome 81
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg
Number analyzed (Participants) | 50 | 55
ng*h/mL | 4.09 (74.3) | 5.52 (61.4)

83. Secondary Outcome: Cumulative Amounts of Ipratropium [μg] Excreted in Urine for 0-2 Hours
Description: Cumulative amounts of Ipratropium [μg] excreted in urine - Planned time intervals 0-2, ss
Time Frame: Before drug administration to 2 hours after drug administration on Day 29
Population: as for outcome 81
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 Mcg
Number analyzed (Participants) | 44 | 51 | 47
μg | 0.747 (148) | 0.692 (180) | 0.723 (220)

84. Secondary Outcome: Cumulative Amounts of Albuterol [μg] Excreted in Urine for 0-2 Hours
Description: Cumulative amounts of Albuterol [μg] excreted in urine - Planned time intervals 0-2,ss.
Time Frame: Before drug administration to 2 hours after drug administration on Day 29
Population: as for outcome 81
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg
Number analyzed (Participants) | 46 | 52
μg | 14.7 (143) | 20.3 (141)

85. Secondary Outcome: Cumulative Amounts of Ipratropium [μg] Excreted in Urine for 0-6 Hours
Description: Cumulative amounts of Ipratropium [μg] excreted in urine - Planned time intervals 0-6,ss
Time Frame: Before drug administration to 6 hours after drug administration on Day 26
Population: as for outcome 81
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Number analyzed (Participants) | 48 | 55 | 51
μg | 1.66 (128) | 1.41 (143) | 1.51 (145)

86. Secondary Outcome: Cumulative Amounts of Albuterol [μg] Excreted in Urine for 0-6 Hours
Description: Cumulative amounts of Albuterol [μg] excreted in urine - Planned time intervals 0-6, ss
Time Frame: Before drug administration to 6 hours after drug administration on Day 29
Population: as for outcome 81
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg
Number analyzed (Participants) | 49 | 55
μg | 33.7 (123) | 39.4 (116)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Serious Adverse Events (participants affected / at risk) | 17 | 33 | 14
Other Adverse Events (participants affected / at risk) | 61 | 51 | 43
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Arteriosclerosis coronary artery (Cardiac disorders) | 0/486 | 1/491 | 0/483
Atrial Fibrillation (Cardiac disorders) | 0/486 | 1/491 | 0/483
Coronary artery disease (Cardiac disorders) | 1/486 | 0/491 | 0/483
Constipation (Gastrointestinal disorders) | 0/486 | 1/491 | 0/483
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0/486 | 1/491 | 0/483
Haemorrhoids (Gastrointestinal disorders) | 0/486 | 1/491 | 0/483
Inguinal hernia (Gastrointestinal disorders) | 0/486 | 1/491 | 0/483
Chest pain (General disorders) | 0/486 | 0/491 | 1/483
Death (General disorders) | 1/486 | 0/491 | 0/483
Oedema peripheral (General disorders) | 0/486 | 0/491 | 1/483
Abscess limb (Infections and infestations) | 1/486 | 0/491 | 0/483
Appendicitis (Infections and infestations) | 1/486 | 0/491 | 0/483
Bronchitis (Infections and infestations) | 3/486 | 2/491 | 0/483
Cellulitis (Infections and infestations) | 1/486 | 0/491 | 0/483
Diverticulitis (Infections and infestations) | 1/486 | 0/491 | 0/483
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1/486 | 1/491 | 0/483
Lobar pneumonia (Infections and infestations) | 0/486 | 2/491 | 1/483
Pneumonia (Infections and infestations) | 2/486 | 3/491 | 3/483
Tracheobronchitis (Infections and infestations) | 1/486 | 0/491 | 0/483
Incisional hernia (Injury, poisoning and procedural complications) | 1/486 | 0/491 | 0/483
Injury (Injury, poisoning and procedural complications) | 0/486 | 1/491 | 0/483
Road traffic accident (Injury, poisoning and procedural complications) | 0/486 | 1/491 | 0/483
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0/486 | 1/491 | 0/483
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/486 | 0/491 | 1/483
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/486 | 1/491 | 0/483
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/486 | 0/491 | 1/483
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/486 | 1/491 | 0/483
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/486 | 1/491 | 0/483
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/486 | 2/491 | 0/483
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/486 | 1/491 | 0/483
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/486 | 0/491 | 1/483
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/486 | 1/491 | 0/483
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/486 | 0/491 | 1/483
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/486 | 0/491 | 0/483
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/486 | 0/491 | 1/483
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/486 | 1/491 | 0/483
Cerebral cyst (Nervous system disorders) | 0/486 | 0/491 | 1/483
Loss of consciousness (Nervous system disorders) | 0/486 | 1/491 | 0/483
Syncope (Nervous system disorders) | 0/486 | 1/491 | 0/483
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0/486 | 1/491 | 0/483
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10/486 | 12/491 | 8/483
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/486 | 2/491 | 0/483
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0/486 | 0/491 | 1/483
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0/486 | 1/491 | 0/483
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0/486 | 0/491 | 1/483
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/486 | 0/491 | 0/483
Angiopathy (Vascular disorders) | 0/486 | 1/491 | 0/483
Thrombophlebitis (Vascular disorders) | 0/486 | 0/491 | 1/483
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | COMBIVENT Respimat 20/100 mcg | COMBIVENT CFC-MDI 36/206 mcg | Ipratropium Respimat 20 mcg
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 61/486 | 51/491 | 43/483

LIMITATIONS AND CAVEATS:
The FEV1 and FVC measurements at each observation time point were used to derive the primary and secondary efficacy endpoints and are not reported here. All statistical analyses for secondary endpoints are exploratory and the p-values are nominal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.